CLINICAL TRIAL: NCT06202352
Title: The Effect of Basic Yoga and Meditation Techniques on Midwifery Students' Anxiety and Perceived Stress Levels
Brief Title: Basic Yoga and Meditation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Funda Citil Canbay, Association Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/585
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Mediation
Keywords: Student; Midwifery; Mediation; Yoga; Stress
MeSH Terms: conditions — Negotiating | interventions — Meditation; Yoga

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The group which yoga and meditation are implemented
  Interventions: Behavioral: Meditation and Yoga
- Control (No Intervention): The group which has no implementation

INTERVENTIONS:
Behavioral: Meditation and Yoga — The yoga and meditation intervention will use a 60-minute vinyasa yoga class once a week, followed by a guided yoga instruction booklet that takes an average of 30 minutes to read. The intervention will be carried out in the last eight weeks of the spring semester, when hospital practices are most intense and before the final exams. Posttest forms will be filled out the week of final exams. The time devoted to meditation will be increased every week for the last two weeks, starting with 5 minutes and gradually increasing to 20 minutes in the eighth week.
  Arms: Intervention Group

SUMMARY:
Purpose of the research; To determine the effect of basic yoga techniques and meditation intervention on midwifery students' anxiety and perceived stress levels.

Yoga is alternative mind-body exercises that aim to establish a connection between the brain and body. Derived from the Sankiritic term "yuj", yoga means to integrate. Yoga techniques focus on self-awareness and require careful coordination of body movements/postures (asanas), deep breathing (pranayama) and meditation. Yoga can be used as a complementary and alternative method for various diseases or improving well-being. Yoga is becoming increasingly important in improving mental health. In this planned study, we aim to manage the anxiety and perceived stress that students studying in the field of health mostly suffer from with yoga techniques.

After the sociodemographic data of the volunteer participants who agree to take part in the research are identified and recorded in the first stage, the screening phase, according to the power analysis, the minimum number of participants determined will be assigned to the experimental and control groups by randomization. In the second stage of the research, the experimental group; Yoga techniques and meditation practices (once a week for 8 weeks) will be performed at times when anxiety and stress are most intense (before exams, laboratory and hospital applications). Students in the control group will continue their routine coping habits with anxiety and stress. Students will complete pre- and post-intervention surveys to assess changes in anxiety and perceived stress. The anxiety and stress levels of students in both groups will be determined by applying the "Beck Anxiety Inventory" and the "Perceived Stress Scale" before and after the intervention. The data obtained after the interventions will be compared with appropriate statistical analysis and converted into a report.

The proposed research aims to provide scientific research skills and experience to the 2nd year students of Atatürk University, Faculty of Health Sciences, Department of Midwifery, who are involved in the project. In addition, it is expected that the proposed project will show how it affects the anxiety and perceived stress levels of midwifery students in the international media and literature and emphasize its positive effects on the management of the well-being of these individuals.

DETAILED DESCRIPTION:
Introduction Derived from the Sanskrit word "yuj", yoga means integrated awareness of mind and body. Yoga techniques are popular practices that include the coordination of different posture techniques, deep breathing practices and meditation (Sarbacker and Kimple, 2015). Since yoga is a mental exercise that slows down brain waves, it can help eliminate negative emotions and ensure awareness and cognitive balance (Desai et al., 2015). It has been understood that controlling perceived stress not only reduces mood disorders, but also provides better sensorimotor performance and hand grip endurance (Bajunaid et al., 2015). Midwifery is a discipline in which theory and practice are carried out in an integrated manner, and it requires the completion of difficult, complex graduation criteria regarding the prenatal, intraparum and postpartum processes (Aydın Kartal and Yazıcı, 2017; Nehir and Güngör Tavşanlı, 2021). In general, in studies conducted on midwifery students, it is observed that stress and anxiety are inevitably high (Aydın Kartal and Yazıcı, 2017; Nehir and Güngör Tavşanlı, 2021). Since today's midwifery students will be the expert midwives of the future, the physical and mental health of midwifery students can increase the welfare of society. In this context, teaching midwifery students to connect with their body and mind may increase psychological well-being.

According to the results of a limited number of studies, yoga exercises provided positive effects on medical/health education students suffering from intense stress and anxiety (Erogul et al., 2014; Fares and Fares, 2016). The limited number of studies conducted in the field of health education on the effects of yoga and meditation focused on students of medicine, pharmacy and nursing departments (Lemay et al., 2019; Ciezar-Andersen et al., 2021). On the other hand, despite the popularity of yoga in studies mostly in western societies (Shohani et al., 2018), to our knowledge, how it prevents mood disorders in the field of midwifery has not been studied. Studies on the effects of yoga are limited in Turkey.

Method The total screening of the project will be carried out in 2 stages. In the first stage, students' anxiety and stress levels will be screened. After the screening study, students' demographic characteristics, general anxiety and perceived stress levels will be measured. According to the data obtained from the scanning study, the numbered forms will be put in order and the data obtained will be recorded in the IBM SPSS (Statistical Package for the Social Sciences) Statistic 21 package program. According to the data obtained as a result of the screening study, participants (72 students) who will be sampled according to their anxiety and perceived stress levels will be assigned to the yoga techniques and control group. A randomization program (www.randomize.org) will be used to assign groups.

Students assigned to groups through randomization will be contacted via their contact numbers and will be informed about the research and which group they will be in. Appointments will be made with students assigned to study groups, and yoga/meditation techniques will begin in a suitable room at the faculty. Meetings will be arranged with the yoga and control groups determined during the selection phase, after the lesson hours of each class. Two separate WhatsApp groups will be created: control and yoga groups. The responsible researcher has an international yoga training certificate.

Yoga and meditation practices (8 weeks, once a week, 60 minutes):

The yoga and meditation intervention will use a 60-minute vinyasa yoga class once a week, followed by a guided yoga instruction booklet that takes an average of 30 minutes to read. The intervention will be carried out in the last eight weeks of the spring semester, when hospital practices are most intense and before the final exams. Posttest forms will be filled out the week of final exams. The time devoted to meditation will be increased every week for the last two weeks, starting with 5 minutes and gradually increasing to 20 minutes in the eighth week.

* Application Place(s) of the Research: It will be carried out in a suitable room at Atatürk University, Faculty of Health Sciences, Department of Midwifery.
* Details of Study Design and Method:

The planned study is a pre-posttest-posttest, randomized controlled experimental study.

• Sample Size Population and Sample of the Research: The population of the study will consist of 724 registered students studying at Atatürk University, Faculty of Health Sciences, Department of Midwifery (1st, 2nd, 3rd, 4th Grade) in the 2023-2024 academic year. The maximum number of students (sample) to be included in the study was calculated using G*Power 3.1.9.7 software. Taking Shohani et al.'s (2018) study titled "The Effect of Yoga on Stress, Anxiety, and Depression in Women" as a reference, it was determined that the effect size of the difference between pre- and post-training individuals in the experimental group who received yoga training was 0.351. Accordingly, the sample size required for 80% (1-β=0.80) power at d = 0, 351 and α = 0.05 was calculated as 33 people from each group. Considering the possibility of midwifery students leaving the groups during the research, it was decided that the number of samples in the groups would be 36, based on a 10% loss. Students who do not meet the inclusion criteria for the study will not be included in the randomization.

Since it is aimed to reach all midwifery students in the survey study, no sample selection will be made. In order to reach eligible students later after the screening, students' contact information will be written in the surveys and the scales will be numbered. At this stage; 72 students who meet the inclusion criteria for this study and volunteer will be divided into control and yoga groups. The dependent variables of the study are yoga and meditation. Independent variables are anxiety level and perceived stress level. Additionally, students will have to sign an Informed Consent Form.

• Collecting Study Data and Recording Data Data Collection Tools Sociodemographic data of midwifery students will be recorded with the "Student Identification and Monitoring Form" prepared by the research team. In addition, the "Beck Anxiety Scale" and "Perceived Stress Scale" will be used for the screening study, before and after the intervention.

Student Diagnosis and Monitoring Form (ANNEX-1) Student Identification and Follow-up Form to be used in collecting research data: A form will be used to inquire about the situations related to name, surname, class, age, height, weight, age, marital status, place of residence, mother and father's working status and attitude towards exercise. This information will be filled in by self-report method.

Beck Anxiety Scale (BAI) (ANNEX-2) The scale evaluates the severity of generalized anxiety symptoms. This instrument focuses on somatic symptoms of anxiety and contains 21 items. Responses are based on a 4-point Likert scale ranging from 0 (not at all) to 3 (severely), with a maximum total score of 63. Scores between 0 and 21 indicate low anxiety, scores between 22 and 35 indicate moderate anxiety, and scores of 36 and above indicate high anxiety. The scale was adapted to the Turkish sample by Durak and Palabıyıkoğlu (Durak and Palabıyıkoğlu, 1994).

Perceived Stress Scale (PSS) (Annex-3) It was adapted into Turkish by Eskin et al. (2013). Measuring stress is important for scientific research and application activities to be carried out in our country. ASÖ reliability coefficient was calculated as 0.87 (Eskin et al., 2013). The scale in question consists of 14 items (Erci, 2006). The scale has two subscales: Perception of Insufficient Self-Efficacy and Perception of Stress/Discomfort; Items 1, 2, 3, 7, 11, 12 and 14 constitute the Perception of Stress/Discomfort dimension, and items 4, 5, 6, 8, 9, 10 and 13 constitute the Perception of Insufficient Self-Efficacy dimension. In the scale, items 4, 5, 6, 7, 9, 10 and 13 are scored reversely. The total score determined as a result of the scale application indicates the stress level. It shows low stress level between 11-26 points, medium stress level between 27-41 points, and high stress level between 42-56 points.

• Application of Research The total screening of the project will be carried out in 2 stages. In the first stage, students' anxiety and stress levels will be screened. After the screening study, students' demographic characteristics, general anxiety and perceived stress levels will be measured. According to the data obtained from the scanning study, the numbered forms will be put in order and the data obtained will be recorded in the IBM SPSS (Statistical Package for the Social Sciences) Statistic 21 package program. According to the data obtained as a result of the screening study, participants (72 students) who will be sampled according to their anxiety and perceived stress levels will be assigned to the yoga techniques and control group. A randomization program (www.randomize.org) will be used to assign groups.

Students assigned to groups through randomization will be contacted via their contact numbers and will be informed about the research and which group they will be in. Appointments will be made with students assigned to study groups, and yoga/meditation techniques will begin in a suitable room at the faculty. Meetings will be arranged with the yoga and control groups determined during the selection phase, after the lesson hours of each class. Two separate WhatsApp groups will be created: control and yoga groups. The responsible researcher has an international yoga training certificate.

* Description of Transactions on Working Days & Visits (if any) Students currently studying at Atatürk University, Faculty of Health Sciences, Department of Midwifery, will be informed about the research and invited to participate in the research. Research data will be collected from students who agree to participate in the research using a survey form and face-to-face interview technique.
* Randomization Method & Importance (if any) Randomization will be provided in an online program. A randomization program (www.randomize.org) will be used to assign groups. Students assigned to groups through randomization will be contacted via their contact numbers and will be informed about the research and which group they will be in.
* Ensuring Patient Compliance (if any) Before starting the research, approval will be obtained from the non-invasive ethics committee of Atatürk University Faculty of Medicine and official permission will be obtained from the Midwifery Department of Atatürk University Faculty of Health Sciences. Midwifery students within the scope of the research will be informed about the research and their informed consent will be obtained before starting to collect research data. In addition, ethical principles including the principle of "confidentiality and protection of confidentiality" will be fulfilled by stating that the information obtained from the students will be kept confidential, and the principle of "respect for autonomy" will be fulfilled by recruiting those who want to participate in the research voluntarily.
* Ensuring volunteer participation and obtaining consent, defining the procedures to be taken in the volunteers' special situations.

Informed voluntary consent, given with the completely free will of the students who will participate in the research, will be obtained from all volunteers before the research is initiated. Information regarding the clinical trial will be recorded in a manner that allows for accurate reporting, interpretation and verification of this information.

* Materials to be Used & Storage Conditions & Responsibilities (if any) Records regarding the identity of volunteers will be protected in a way that respects the rules of private life and confidentiality in accordance with the relevant legislation. Survey forms will be kept by the principal investigator for at least five years.
* Statistical & Analytical Methods should be clearly stated in this section. After yoga practices are completed, post-test forms (Perceived Stress Scale and Beck Anxiety Scale) will be administered. The data obtained as a result of the study will be recorded in the IBM SPSS (Statistical Package for the Social Sciences) Statistic 21 package program and statistical analysis will be performed.

First of all, Kolmogorov-Smirnov Goodness of Fit Test and "Shapiro-Wilk" will be applied for normality analysis in determining the test to be performed. In descriptive statistics, arithmetic mean, standard deviation, median, minimum and maximum values will be applied, and frequency and percentage will be applied to categorical variables. Cronbach's Alpha Coefficient will be calculated to test the internal consistency of the scales. "Pearson Chi-square Test and Fisher's Exact Test" will be applied to compare the descriptive characteristics between the study and control groups. Within-group paired sample t -test to compare pre- and post-intervention results, based on established normality.

(Paired-Samples T test) will be applied. In determining the difference between the two group averages, t-test will be applied in independent groups. The statistical significance level will be accepted as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have the skills and competence to do Vinyasa yoga exercises,
* Having no obstacle to exercise,
* Does not have any chronic disease,
* Students who have not received yoga training before and are not pregnant.
* Those who do not have any symptoms that may be related to breathing or heart rhythm,
* Having no orthopedic and/or neurological sequelae that prevent exercise,
* Volunteer and willing participants will be included.

Exclusion Criteria:

* Those whose vital and health conditions are unstable
* Disability
* Those who have a diagnosed psychological disease and are using active medication
* Students with harmful habits such as smoking and alcohol will not be included in the scope of the research.
* Students who are not willing to participate in the research, fill out the research forms incompletely, and have communication problems will be excluded from the scope of the research.
* Students who do not want to continue the research will be excluded from the research.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | 12 months
  The effect of yoga and meditation on anxiety
Stress Perception | 12 months
  The effect of yoga and meditation on stress perception

CONTACTS AND LOCATIONS:
Locations (1):
- Funda Çitil Canbay, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want to provide information about plans to share individual participant data (IPD).